CLINICAL TRIAL: NCT05685056
Title: Nutrition and Food Choices in Early Pregnancy - a Nutrition Education Intervention
Brief Title: Nutrition & Food Choices in Early Pregnancy
Acronym: PICk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Glasgow (Other)
Responsible Party: Principal Investigator, Emilie Combet, Principal Investigator, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 200160090
Record Dates: First submitted 2017-10-30; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Iodine Deficiency
Keywords: Iodine; Pregnancy; Food choices; Fish; Dairy

STUDY DESIGN:
Who Masked: Participant
Masking Description: Both groups (control and intervention) will be informed that the main aim of the study is to assess the impact of food guidance on the micronutrient intake in pregnant women. The intervention group will receive texts with detailed information focusing on nutrition and iodine rich foods specifically. The information sheet will have information on all the study procedures but the focus on iodine will remain discreet, to avoid unintended bias in response from participants. At the end of the study, participants will be debriefed on the deception.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group will receive no intervention, and will be receiving only text reminders regarding the study, the following visits and study logistics in order to limit dropout rate.
- Intervention group (Experimental): Intervention will happen with weekly text messages during the study period, focusing on pregnancy nutrition and iodine rich foods. The texts will be based on the taxonomy of behavior change techniques used in interventions, the nudge theory and will be covering themes identified on our previous research.
  Interventions: Behavioral: Text messages

INTERVENTIONS:
Behavioral: Text messages — Texts with detailed information focusing on nutrition and iodine rich foods specifically, every 3-5 days.
  Arms: Intervention group

SUMMARY:
PICk study is a mHealth intervention in women trying to conceive and women up to 14 weeks pregnant, aiming to guide food choices, to achieve the recommended iodine intake through diet.

DETAILED DESCRIPTION:
Iodine is important for the synthesis of thyroid hormones, which are driving normal brain development in fetal and postnatal life.

The required level of iodine intake is 140μg/day and there is not proposed increment for pregnant women from the United Kingdom (UK) Department of Health, in contrast to the World Health Organisation (WHO), EFSA, US Institute of Medicine (IoM) and SANZ, that propose an intake in pregnancy which varies from 200 to 150μg/day. In the UK, based on our previous findings, 60% of women in pregnancy do not meet the 250μg/day WHO recommendation of intake.

Over half mothers and practitioners in the UK were found to be unable to identify correct sources of iodine. However, most women have reported willingness to modify dietary behaviour if they received information related to the importance of iodine in pregnancy.

This intervention focuses on providing information about iodine and its importance in pregnancy that would potentially help women improve their iodine status. The intervention was designed with participants involvement and their views on best way of getting information, informed by in-depth qualitative work.

The hypothesis is that increasing knowledge and awareness about the importance, sources and requirements of iodine during pregnancy will lead to change in practice and increased iodine intake.

Methods:

The study is a randomised controlled trial that lasts for 12 weeks. Women in preconception and in the 1st pregnancy trimester will be recruited and will be randomised either to the control or to the intervention group.

The study involves 3 meeting with the participants, at baseline and after 6 and 12 weeks. For women who try to conceive, if conception occurs within the study period, there is a fourth (optional) meeting in the 12th week of pregnancy.

Participants are informed about the study without getting details of the aim (to increase the iodine status of those in the treatment group). This is in order to decrease any bias and avoid leading participants to self-research the topic of iodine nutrition. Women of both study arms receive standard care and the study will not aim to change this. The treatment group is to receive 1-2 weekly text messages focusing on iodine-rich foods importance, barriers identification and tips with ways to include them in the diet.

Samples collection and analysis:

* Questionnaires (demographic, dietary, knowledge, awareness and intervention assessment questionnaires) will be completed by the participants at the place of recruitment / meeting with the researcher after full instructions by the researcher in visits 1, 2 and 3 (and optional visit 4).
* Participants will be given 12 pots for spot urine samples collection in each visit. They will be asked to collect 10 urine samples over 3-4 days. Urinary iodine and creatinine concentrations will be measured.
* A finger prick dried blood spot sample will be taken from each participant in each visit by the researcher. Thyroglobulin will be measured.

Power calculation:

The primary aim of the study is to decrease the proportion of women not meeting the recommended intake for iodine.

Based on a proportion of 60% of women currently not meeting the 250 μg/day recommended intake 5, a sample size of N=84 in total (42 per group) would allow to detect a decrease in proportion down to 30%. This is achievable based on the % of women with an intake of 150-249 μg/day, who could increase consumption by 100 μg/day (equivalent to a 200ml portion of milk and a 125g portion of yoghurt per day) and therefore meet the threshold. Adjusting for 15% dropout, a sample of 50 per group would be sufficient.

ELIGIBILITY:
Inclusion Criteria:

* Trying to conceive or first trimester pregnant women
* English speaking
* Healthy

Exclusion Criteria:

* Abnormal pregnancies
* Known thyroid disorders, renal disease, multiple pregnancies, development of gestational diabetes
* Participation in another trial
* Not owning a mobile phone
* Followed by a dietitian at the time of the trial
* Existing or past eating disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female because pregnancy focus
Enrollment: 100 (Actual)
Dates: Start 2017-03-25 (Actual); Primary Completion 2019-06-17 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
proportion of women not meeting the recommended intake for iodine | 6 weeks
  measured by validated food frequency questionnaire
proportion of women not meeting the recommended intake for iodine | 12 weeks
  measured by validated food frequency questionnaire

SECONDARY OUTCOMES:
iodine awareness | 6 weeks
  Measured by questionnaire, as a median score
iodine awareness | 12 weeks
  Measured by questionnaire, as a median score
Iodine knowledge | 6 weeks
  Measured by questionnaires, as a median score
Iodine knowledge | 12 weeks
  Measured by questionnaires, as a median score
Thyroglobulin concentration | 6 weeks
  measured by immunoassay
Thyroglobulin concentration | 12 weeks
  measured by immunoassay
Change in urinary iodine concentration (from baseline) | 6 weeks
  measured by colorimetry
Change in urinary iodine concentration (from baseline) | 12 weeks
  measured by colorimetry

CONTACTS AND LOCATIONS:
Locations (1):
- Community, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided